CLINICAL TRIAL: NCT02441816
Title: VITAL - Individualising Therapy for Neovascular AMD With Aflibercept
Acronym: VITAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-002381-73
Record Dates: First submitted 2014-10-20; First posted 2015-05-12 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Age Related Macular Degeneration
Keywords: wet AMD; neovascular AMD
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eylea Treatment (Other): The intravitreal dose of Eylea will be 2mg (in 0.05ml) per injection. The medication will be supplied in single use vials. Given monthly for 3 months and then every 8 weeks in the first year of treatment before applying a treat and extend paradigm to patient visits in year 2. This is an open-label study.
  Interventions: Drug: Aflibercept; Other: Extend Treatment

INTERVENTIONS:
Drug: Aflibercept
  Other Names: Eylea
Other: Extend Treatment — In year 2 of the study a treat and extend protocol will be applied, if a patient has signs of disease activity (eg macular fluid on SDOCT) they will be brought back at 8 weeks after the visit and given an intravitreous injection. They will then be reviewed 8 weeks post treatment for a further treatment with follow-up and treatment interval extended to 10 weeks if the disease is quiescent (if no macular fluid at the subsequent visit the patient could be extended to 12 weeks interval with treatment).

SUMMARY:
The purpose of this study is to assess a new treatment pattern for aflibercept. The aim is to achieve and maintain the best benefit of visual function and avoid unnecessary hospital visits.

The hypothesis to be tested is whether intravitreous aflibercept given in an 8 week cycle of treatment in year 1 and a capped treat and extend treatment paradigm in year 2 can lead to improved vision and reading speed in eyes with active wet AMD over 2 years while reducing hospital visits.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥ 50 years of either gender
* Women must be postmenopausal for at least 12 months prior to trial entry, or surgically sterile. If of child bearing potential, a serum pregnancy test with a negative result must be obtained within 14 days prior to the first treatment.
* Women of child bearing potential must be practicing effective contraception implemented during the trial and for at least 60 days following the last dose of study medication.
* No condition that precludes follow-up for 2 years.
* No contraindication to intravitreous injection of aflibercept.

Study eyes must meet the following criteria for entry into the trial and must have vision loss accounted for by wet AMD:

* Newly diagnosed, angiographically documented, previously untreated, active CNV lesion (i.e., leakage on fluorescein angiography AND subretinal, intraretinal, or sub-RPE fluid on OCT) secondary to age-related macular degeneration.
* Best corrected visual acuity score in the study eye of between 80 and 23 letters inclusive, using ETDRS testing, (between 6/7.5 and 6/96 Snellen equivalent), inclusive.
* The CNV or sequela of the CNV (i.e., pigment epithelium detachment, subretinal haemorrhage, blocked fluorescence, macular edema, or subretinal or intraretinal fluid) must involve the centre of the fovea.
* The total area of fibrosis must comprise less than 50% of the total lesion.
* > 1 drusen (>63 microns) in either eye OR late AMD in fellow eye
* No previous treatment for CNV in the study eye
* Clear ocular media and adequate pupillary dilation to permit good quality fundus imaging.

Exclusion Criteria:

Subjects who meet the following criteria will be excluded from study participation:

6.2.1 Prior/Concomitant Treatment

* Any previous treatments for wet AMD (including verteporfin PDT, Macugen®, Lucentis®, intravitreous Avastin®, thermal laser, external beam radiation or surgery for AMD) in the study eye
* Current or planned use of systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/ hydroxychloroquine (Plaquenil®), phenothiazines and ethambutol.
* Previous participation in any studies of investigational drugs likely to have ocular effects within 30 days preceding the initial study treatment
* Concurrent or previous use of systemic anti-VEGF agents.
* Any intraocular procedure (including Yttrium-Aluminium-Garnet capsulotomy) within 2 months prior to Screening or anticipated within the next 6 months following Screening 6.2.2 Lesion Characteristics
* Permanent structural damage (fibrosis or atrophy) involving the centre of the fovea in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelial tear involving the fovea in the study eye 6.2.3 Concurrent Ocular Conditions
* Any concurrent intraocular condition in either eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either require medical or surgical intervention during the 2 year follow-up period to prevent or treat visual loss that might result from that condition, or, if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 2 year follow-up period.
* Active or recent (within 4 weeks) intraocular inflammation (grade trace or above) in either eye
* Neovascularisation of the iris, neovascular glaucoma or vitreous haemorrhage in either eye at the screening visit
* History of rhegmatogenous retinal detachment, epiretinal membrane, vitreomacular traction or macular hole in the study eye if in the investigators opinion, thought to limit potential for vision improvement after treatment for wet AMD
* History of vitrectomy in study eye
* Active infectious conjunctivitis, blepharitis, keratitis, scleritis, or endophthalmitis in either eye at the time of screening
* Spherical equivalent of the refractive error in the study eye demonstrating more than 8 diopters of myopia
* For subjects who have undergone prior refractive or cataract surgery in the study eye, the preoperative refractive error in the study eye cannot exceed 8 diopters of myopia.
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding the first study treatment.
* Uncontrolled glaucoma in either eye at the time of screening (defined as intraocular pressure >25 mmHg despite treatment with anti-glaucoma medication)
* Inability to be photographed or to document CNV (eg due to allergy to fluorescein dye, lack of venous access or cataract obscuring the CNV).
* Inability to obtain OCT images of reasonable quality to allow analysis of lesion or macular fluid
* Patients with other ocular diseases or conditions that can compromise the visual acuity of the study eye such as amblyopia, anterior ischemic optic neuropathy, previous complicated cataract surgery, aphakia, vitreomacular traction or diabetic macular oedema 6.2.4 Concurrent Systemic Conditions
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation. Females of childbearing potential must have a negative pregnancy test within 14 days prior to being registered for trial treatment NOTE: Subjects are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Pregnancy or breastfeeding
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
* History of recurrent significant infections or bacterial infections
* Inability to comply with study or follow-up procedures
* Stroke or myocardial infarction less than 3 months from Screening date
* Known hypersensitivity to aflibercept

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Primary outcome - mean change in visual acuity (Early Treatment of Diabetic Retinopathy Study letter score) | 24 months
  The primary outcome is the mean change in visual acuity (Early Treatment of Diabetic Retinopathy Study letter score) at 24 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Patel, MD, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Patel PJ, Jayaram H, Eleftheriadou M, Vazquez-Alfageme C, Islam N, Rubin GS, Pal B, Addison PK, Hamilton R, Degli Esposti S. Individualizing Therapy for Neovascular Age-Related Macular Degeneration with Aflibercept (VITAL): A Two-Year Prospective, Interventional Single-Centre Trial. Ophthalmol Ther. 2020 Sep;9(3):563-576. doi: 10.1007/s40123-020-00267-5. Epub 2020 Jun 18. PMID 32557168